CLINICAL TRIAL: NCT06708065
Title: Outcomes of Combining Armeo Power Robotic Therapy with Conventional Rehabilitation for Upper Limb Motor Recovery in Patients with Hemiplegia Following Supratentorial Cerebral Infarction
Brief Title: Effects of Armeo Power Robot Therapy on Upper Limb Recovery in Hemiplegic Stroke Patients
Acronym: BV108/RAPPHCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: The 108 Military Central Hospital (Other Government)
Responsible Party: Principal Investigator, Tuan Nguyen Thanh, Dr, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1139/GCN-HMUIRB
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Rehabilitation of Upper Limb Motor Function in Hemiplegia Due to Supratentorial Cerebral Infarction Using Armeo Power Robot
Keywords: robot Armeo Power, upper extremity function, rehabilitation, ischemic stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: 1. 84 hemiplegic patients, diagnosed with supratentorial cerebral infarction, were treated for stable stroke at clinical departments, meeting the inclusion and exclusion criteria.
  2. Dividing the intervention group and the control group according to the lottery method of sampling.
  3. Intervention content:
     * Control group: 42 patients were assigned to: regular physical therapy and occupational therapy, 90 minutes/day x 5 days/week. In addition, patients were instructed to practice at home 45 minutes/day x 5 days per week (direct instruction combined with distributing leaflets of exercises).
     * Intervention group: 42 patients were assigned to: regular physical therapy and occupational therapy, 90 minutes/day x 5 days/week. In addition, patients were trained with the Armeo Power robot 45 minutes/day, 5 days per week. - The research subjects were examined and evaluated at two points in time:
     * Time 1: Before intervention
     * Time 2: After completing 3 weeks of training (15 sessions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ARMEO group (Experimental): The intervention group consisted of 42 patients who received standard physical therapy and occupational therapy for 90 minutes per day, five days per week. Additionally, these patients underwent training with the ArmeoPower robotic system for 45 minutes per day, five days per week.
  Interventions: Device: Armeo Power robot restores upper limb motor function.; Behavioral: A Home Exercise Program; Behavioral: Occupational therapy activities
- Control group (Active Comparator): The control group comprised 42 patients who participated in standard physical therapy and occupational therapy for 90 minutes per day, five days per week. In addition, these patients were instructed to engage in home-based practice for 45 minutes per day, five days per week, guided by direct instructions and exercise leaflets provided by the therapists.
  Interventions: Behavioral: A Home Exercise Program; Behavioral: Occupational therapy activities

INTERVENTIONS:
Device: Armeo Power robot restores upper limb motor function. — ArmeoPower is a robotic rehabilitation device developed by Hocoma, designed to assist patients with impaired upper limb motor functions following conditions such as stroke or neurological injuries. The device features an exoskeleton that supports and tracks movements of the arm and hand, utilizing motor-assisted motion based on the principle of "adaptive support," which adjusts assistance levels according to the patient's capabilities. ArmeoPower integrates interactive exercises, often in the form of engaging games, to enhance patient motivation and maintain focus during therapy sessions. It also collects and tracks performance data, enabling clinicians to evaluate progress over time. This device is widely used in rehabilitation centers and hospitals to improve muscle control, strength, and range of motion in patients recovering from severe motor impairments.
  Arms: ARMEO group
Behavioral: A Home Exercise Program — A Home Exercise Program (HEP) is a personalized set of exercises designed to support recovery and enhance functional abilities outside of clinical therapy sessions. For patients with hemiplegia due to cerebral infarction, the program typically includes range of motion (ROM) exercises to maintain joint flexibility and prevent stiffness, as well as strengthening exercises using resistance bands or light weights to improve muscle function. Balance and postural control exercises, such as weight shifting or standing on one leg, help enhance stability and reduce fall risks. Functional training focuses on practicing daily movements like reaching, grasping, or transferring between positions, while fine motor skill tasks aim to restore hand functionality. The program may also incorporate low-impact aerobic exercises, such as walking or seated cycling, to boost cardiovascular health, along with relaxation and breathing techniques to reduce stress and improve overall well-being. These exercises a
Behavioral: Occupational therapy activities — Occupational therapy activities are designed to help individuals regain independence in daily life by addressing functional abilities, motor skills, and cognitive functions. For patients with hemiplegia due to cerebral infarction, these activities often include practicing Activities of Daily Living (ADLs) such as dressing, grooming, bathing, and feeding, as well as more complex tasks like cooking and managing finances. Fine motor skills development is emphasized through exercises involving tasks like buttoning, tying shoelaces, or handling small objects, sometimes using adaptive tools. Additionally, functional mobility training focuses on teaching safe movement strategies, such as transferring between surfaces or navigating stairs, and may include wheelchair mobility or energy conservation techniques. These activities are tailored to the patient's needs to enhance their ability to perform meaningful and necessary daily tasks independently.

SUMMARY:
This study investigates the effectiveness of combining Armeo Power robotic therapy with conventional rehabilitation techniques to improve upper limb motor function in patients with hemiplegia caused by supratentorial cerebral infarction (a type of stroke). The study aims to evaluate how robotic-assisted therapy can enhance recovery by measuring motor function improvements over three weeks of treatment. Participants will undergo standard physical and occupational therapy alongside Armeo Power training, with results compared to those receiving only standard rehabilitation. The findings aim to provide valuable insights into advanced therapeutic options for stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria

* Spasticity of the affected arm with a Modified Ashworth Scale score ≤ 2.
* Patients must have good cognition and awareness (MoCA score ≥ 26).
* Patients must have good vision and visual perception.
* Patients must have stable sitting posture and good sitting balance.
* Body weight and affected arm size must be compatible with the robotic arm device.
* Patients must agree to participate in the study and adhere to the training protocol.

Exclusion Criteria

* Spasticity with a Modified Ashworth Scale score ≥ 3.
* Severe sensory impairment in the affected limb.
* Patients with arthritis or joint stiffness.
* Hemiplegia caused by conditions other than stroke.
* Pre-existing motor disabilities in the affected limb before the stroke.
* Skin lesions on the limb requiring rehabilitation.
* Uncontrolled epilepsy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Comparison of upper limb motor function improvement according to 3 scales: FMA-UE, ARAT and HMS in 2 study groups. | There are 2 time points for evaluating the research subjects in both groups: Time 1: before intervention Time 2: After the end of 15 intervention sessions (about 3 weeks)
  The Fugl-Meyer Assessment for Upper Extremity (FMA-UE) is a standardized clinical test used to evaluate the recovery of upper limb motor function in patients after a stroke. This scale is widely recognized for its reliability and sensitivity in assessing motor recovery during rehabilitation. The test comprises 8 assessment domains with a total of 33 items, and the maximum score achievable is 66 points. Based on the total score, recovery is categorized into four levels: good (56-66 points), indicating near-complete recovery of motor function; fair (42-54 points), reflecting moderate recovery; average (22-40 points), representing limited recovery with partial functionality; and poor (0-20 points), signifying severe motor impairment

SECONDARY OUTCOMES:
Action Research Arm Test | The Action Research Arm Test (ARAT) can be administered at two time points: baseline (initial assessment) and after 3 weeks to evaluate changes in upper limb function over the course of rehabilitation.
  The Action Research Arm Test (ARAT) is a clinical scale designed to assess upper limb function, encompassing both gross motor skills and fine motor skills of the hand and fingers. The test evaluates four primary categories of movement: grasping large objects, grasping medium-sized objects, pinching small objects, and gross arm movements. The maximum score for the ARAT is 57 points, with recovery outcomes classified into three levels: good recovery (57 points), indicating full restoration of function; moderate recovery (10-56 points), reflecting partial functional ability; and poor recovery (<10 points), signifying severe impairment.
Hand Movement scale | can be administered at two time points: baseline (initial assessment) and after 3 weeks to evaluate changes in upper limb function over the course of rehabilitation.
  The Hand Movement Scale (HMS) is a clinical tool used to evaluate the motor function of the hand and fingers. The scale is divided into six levels, with scores ranging from 1 to 6, corresponding to increasing levels of movement and dexterity. The scoring reflects progression from no movement (1 point) to the highest level, which is the ability to oppose the thumb (digit I) to the other fingers (6 points). The HMS results are categorized into two levels: poor function (1-3 points) and good function (4-6 points)

CONTACTS AND LOCATIONS:
Locations (1):
- 108 Military Central Hospital, Hanoi, Hanoi, Vietnam